CLINICAL TRIAL: NCT01743313
Title: Hyperglycemia in Joint Replacement Recipients: Glucose Metabolism Disorders and Metabolic Syndrome in Osteoarthritis Patients Before and After Primary Hip and Knee Replacement
Brief Title: Glucose Metabolism Disorders and Metabolic Syndrome Before and After Primary Hip and Knee Replacement
Acronym: HyTe-2
Status: Terminated | Type: Observational
Why Stopped: Primary researcher not able to continue research at the moment.
Sponsor: Coxa, Hospital for Joint Replacement (Other)
Collaborators: Tampere University (Other); Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Esa Jamsen, MD, PhD, Researcher, Coxa, Hospital for Joint Replacement
Other Study IDs: HyTe-2
Record Dates: First submitted 2012-12-02; First posted 2012-12-06 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Hyperglycemia; Hypercholesterolemia; Persistent Postoperative Pain; Hip Replacement; Knee Replacement
Keywords: glucose metabolism disorders; metabolic syndrome; joint replacement; osteoarthritis
MeSH Terms: conditions — Hyperglycemia; Hypercholesterolemia; Glucose Metabolism Disorders; Metabolic Syndrome; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples (one per patient).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hip and knee replacement recipients: Hip and knee replacement recipients (with osteoarthritis) enrolled previously into "Perioperative Hyperglycaemia in Primary Total Hip and Knee Replacement" study (NCT01021826).

SUMMARY:
Osteoarthritis patients undergoing primary hip and knee replacement are followed-up and changes in their glucose metabolism and other metabolic parameters (obesity, cholesterol levels) are examined. Persistent postoperative pain is examined as secondary outcome.

DETAILED DESCRIPTION:
Glucose metabolism disorders (diabetes and pre-diabetes) and metabolic syndrome are common in joint replacement recipients. Improved physical activity following joint replacement could lead to better glucose control in diabetes and ameliorate impaired glucose and cholesterol levels. In this study patients previously recruited to "Perioperative Hyperglycaemia in Primary Total Hip and Knee Replacement" study are being followed-up for one year in order to analyze if joint replacements have an effect on these metabolic abnormalities. In addition, the effect of glucose metabolism disorders on occurrence of persistent pain after surgery is analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip and knee replacement for osteoarthritis
* Enrolled previously into study NCT01021826

Exclusion Criteria:

* Arthritis other than osteoarthritis (based on study NCT01021826)
* Medication affecting glucose metabolism (excl. antidiabetic agents) (based on study NTC01021826)
* Died before follow-up phase
* Did not undergo the planned hip or knee replacement

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in glucose tolerance, measured using oral glucose tolerance test | Baseline and 12-24 months after surgery
  The patients are grouped into three groups that are evaluated 12, 18 and ca. 24 months after surgery.

SECONDARY OUTCOMES:
Change in cholesterol levels (HDL, LDL, triglycerides) | Baseline and 12-24 months after surgery
Prolonged postoperative pain | 12-24 months after surgery
  Assessed using visual analog scale. Patients are divided in three groups that are evaluated 12, 18 and 24 months after surgery.

OTHER OUTCOMES:
Change in plasma adipokine and cytokine concentrations | Baseline and 12-24 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Esa Jämsen, MD, PhD, Study Director — Coxa, Hospital for Joint Replacement
Locations (1):
- Coxa, Hospital for Joint Replacement, Tampere, Finland

REFERENCES:
- [Result] Rajamaki TJ, Jamsen E, Puolakka PA, Nevalainen PI, Moilanen T. Diabetes is associated with persistent pain after hip and knee replacement. Acta Orthop. 2015;86(5):586-93. doi: 10.3109/17453674.2015.1044389. PMID 25953426